CLINICAL TRIAL: NCT05481229
Title: Nutritional Status of Cured Pediatric Cancer Patients in Adulthood, the Role of Adipokines in the Development of Cardiometabolic Complications and Desirable Nutritional Interventions
Brief Title: Nutrition Childhood Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: NUTRICE CCS BRNO 2017
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Childhood Cancer; Nutrition Disorders
Keywords: children cancer survivors; adiposity; late effects; nutriton; adipokines
MeSH Terms: conditions — Neoplasms; Nutrition Disorders; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will undergo analysis of peripheral blood (serum or plasma) or urine including characterization of adipokine profiles/metabolites by targeted or untargeted proteomic approach using mass spectrometry (NanoLC/ESI LTQ-Orbitrap MS/MS) or immunoassays (LUMINEX, ELISA) to identify approximately 15-20 molecules associated with cardiometabolic risk;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nutritional interventions — Nutritional intervention will be initiated in patients at risk of overweight and obesity. A targeted nutritional intervention will be carried out, which will include consultation on dietary habits and physical activity as determined by diet and physical activity records. Consultations will be aimed at improving lifestyle and maintaining an adequate body weight.

SUMMARY:
NUTRITION CCS is a cross-sectional, descriptive study to assess the relationship between body composition and demographic, socioeconomic status, treatment modalities and blood samples of survivors who were in remission. The study was conducted in the Clinic for childhood cancer survivors. The clinic is attended by patients older than 18 years and was built in 2016 at the St. Anne's Hospital in Brno.

DETAILED DESCRIPTION:
NUTRITION CCS is a cross-sectional, descriptive study to assess the relationship between body composition and demographic, socioeconomic status, treatment modalities and blood samples of survivors who were in remission.

Objectives of the study

1. to determine the prevalence (incidence) of nutritional disorders, especially obesity and metabolic syndrome, in cured paediatric cancer patients in adulthood;
2. to investigate the role of adipokines in the development of cardiometabolic complications in this group of patients; 3. to determine whether targeted dietary and lifestyle interventions can lead to improvements in nutritional status and subjectively perceived quality of life of treated paediatric cancer patients in adulthood and objectively assessed cardiometabolic risk

ELIGIBILITY:
Inclusion Criteria:

* Patients after treatment from childhood and adolescent cancers.
* The subject is male or female, aged 18 - 64 years

Exclusion Criteria:

* Patients with acute cancer therapy
* Pregnant women

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is patients who have been treated for childhood or adolescent cancer and who are now being followed up in a dispensary clinic.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2023-04-25 (Estimated); Study Completion 2023-04-25 (Estimated)

PRIMARY OUTCOMES:
Define the relationship between the levels of adipokines and cardiometabolic diseases. | through study completion, an average of 1 year
  Define the relationship between the levels of selected adipokines and the risk of selected chronic diseases, specifically cardiometabolic diseases.

SECONDARY OUTCOMES:
Determine the prevalence of hight body fat and decreased skeletal muscle. | through study completion, an average of 1 year
  Determine the number of patients with a high body fat percentage. In these patients, monitor the responses of selected adipokine levels to targeted nutritional intervention leading to fat mass reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bienertová-Vašků, Prof., Principal Investigator — Department of Pathological Physiology and RECETOX, Masaryk University, Kamenice 5,
Locations (2):
- Czechia (2):
  - Masaryk University, Brno
  - St. Anne Hospital in Brno, Brno

REFERENCES:
- [Derived] Strublova L, Kepak T, Kuruczova D, Zlamal F, Holikova M, Kepakova K, Sterba J, Bienertova-Vasku J. Socioeconomic status and adiposity in childhood cancer survivors: A cross-sectional retrospective study. PLoS One. 2024 Feb 16;19(2):e0298068. doi: 10.1371/journal.pone.0298068. eCollection 2024. PMID 38363727